CLINICAL TRIAL: NCT05338125
Title: Identification of the Posterior Lobe of the Human Pituitary Gland During Surgery Using Its Electrophysiological, Neural Signature
Brief Title: Electrophysiology of the Human Pituitary Gland
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too busy for recruitment
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, wrvanfurth, MD, PhD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P19.032
Record Dates: First submitted 2021-11-03; First posted 2022-04-20 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Pituitary Adenoma; Pituitary Tumor; Diabetes Insipidus Cranial Type; Endocrine; Deficiency
Keywords: Electrophysiology
MeSH Terms: conditions — Pituitary Neoplasms; Diabetes Insipidus, Neurogenic

STUDY DESIGN:
Intervention Model Description: Pilot proof-of-concept study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Patients undergoing the extra intra-operative electrophysiological measurement
  Interventions: Procedure: Micro-electrode measurement

INTERVENTIONS:
Procedure: Micro-electrode measurement — Electrophysiological measurement with single-unit micro-electrode

SUMMARY:
Measurment of electrophysiological properties of the human pituitary gland during removal of a pituitary adenoma. Assessment if these properties are sufficient for intra-operative identification of different tissues.

DETAILED DESCRIPTION:
In this study, patients undergoing a surgical resection of a pituitary adenoma as part of standard care will undergo an extra measurement of the electrophysiological properties of the pituitary gland. A single-unit microlectrode will be introduced and placed in the adenoma tissue, anterior piuitary lobe and posterior pituitary lobe. Apart from this measurement, no other interventions are performed and standard care will continue. Six months after measurements the patients chart will be assessed for the occurrence of remission and endocrine deficiencies.

An assessment will be made if these properties are distinctive enough to allow intra-operative identification of the different tissues and thereby increase chances of maximal tumour removal and decrease chance of endocrine deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients undergoing transsphenoidal surgery for pituitary adenoma.
* Identification of the posterior lobe on preoperative MRI. This is most common in patients with micro-adenomas or small macroadenomas.
* Age >18 years

Exclusion Criteria:

* Emergency surgery
* Cognitive impairments
* Pregnancy
* Pre-existing diabetes insipidus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Electrophysiological properties | Day 0
  Electrophysiological properties of the human pituitary gland

SECONDARY OUTCOMES:
Endocrine remission | 6 months postoperative
  Occurrence of endocrine remission after surgery
Endocrine deficiencies | 6 months postoperative
  Occurrence of endocrine deficiencies after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided